CLINICAL TRIAL: NCT05059886
Title: The Injury and Its Consequences in the Sports Lower Limb Amputee
Acronym: PREV'AMP SPORT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2021/GM-01; 2021-A01657-34 (Registry Identifier: ID-RCB (ANSM))
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Leg Lower Amputation; Traumatic Amputation
Keywords: sport; lower limb amputation
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lower limb amputee: No intervention, pure observational study
  Interventions: Other: completion of a questionnaire on the practice of sports and possible injuries

INTERVENTIONS:
Other: completion of a questionnaire on the practice of sports and possible injuries — completion of a questionnaire on the practice of sports and possible injuries

SUMMARY:
This study was motivated by the lack of data in the literature on the injury of the major lower limb amputee playing sports and its socio-professional impact.

It aims to study sports-related injuries in lower limb amputees. Its objective is to determine the prevalence, but also to describe the injuries (type, location, duration, type of management) and their repercussions in terms of after-effects, and repercussions on sports, professional and personal practice. It also aims to begin a correlation between injury and sports load, type of sport (discipline, practice modality), technical aids used

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputee or lower limb agenes
* Amputee before 55 years old
* Amputee for more than 2 years
* Willing to participate in the study
* Practicing a regular physical activity (at least 1x/week)
* Patient affiliated or beneficiary of a health insurance plan.
* Patient aged 18-65 years

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower limb amputee or agenic lower limb with regular physical activity (at least 1x/week)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
prevalence of injuries | in the 5 years preceding the completion of the questionnaire
  presence of injuries (Yes/No, if yes, Nb)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No